CLINICAL TRIAL: NCT03881319
Title: The Study of Efficacy and Effect of Different Dose Acupuncture on Autonomic Nervous Activity and Quality of Life in Women With Dysmenorrhea
Brief Title: The Efficacy of Different Doses of Acupuncture in Dysmenorrhea
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Taipei City Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TCHIRB-10701111
Record Dates: First submitted 2018-11-01; First posted 2019-03-19 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2018-07

CONDITIONS: Premenstrual Syndrome; Dysmenorrhea
Keywords: Acupuncture; Premenstrual Syndrome; Dysmenorrhea; Autonomic nervous activity; TCM syndrome; Meridian
MeSH Terms: conditions — Premenstrual Syndrome; Dysmenorrhea | interventions — Anti-Inflammatory Agents, Non-Steroidal; Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conventional Gynecologic Treatment group (Active Comparator): Taking NSAIDs or oral contraceptives.NSAIDs include Ibuprofen, Naproxen, Diclofenac, and Piroxicam. Oral contraceptives include Yasmin.
  Interventions: Drug: Conventional gynecologic treatment
- Low dose acupuncture group (Experimental): Acupuncture has fewer acupuncture points.
  Interventions: Device: Low dose acupuncture
- High dose acupuncture group (Experimental): Acupuncture has more acupuncture points.
  Interventions: Device: High dose acupuncture

INTERVENTIONS:
Drug: Conventional gynecologic treatment — Taking NSAIDs or oral contraceptives.NSAIDs include Ibuprofen, Naproxen, Diclofenac, and Piroxicam. Oral contraceptives include Yasmin.
  Other Names: NSAIDs or oral contraceptives treatment
  Arms: Conventional Gynecologic Treatment group
Device: Low dose acupuncture — Six acupoints: Three Yin Intersection( SP6)、Grandfather Grandson(SP4)、 Sea of Blood(SP10) 、Sea of Qi(RN6)、Origin Pass(RN4) 、Inner Pass(PC6)
  Arms: Low dose acupuncture group
Device: High dose acupuncture — Twelve acupoints: Three Yin Intersection( SP6)、Grandfather Grandson(SP4)、 Sea of Blood(SP10) 、Sea of Qi(RN6)、Origin Pass(RN4) 、Middle Extremity(RN3)、Inner Pass(PC6) 、Supreme Rush(LR3) 、Joining Valley(LI4) 、Supreme Stream(KI3) 、Uterus(EX-CA1) 、Leg Three Miles(ST36)
  Arms: High dose acupuncture group

SUMMARY:
Subjects in this study included premenstrual syndrome and dysmenorrhea.

Premenstrual syndrome (PMS) is the sum of a group of symptoms (including physical and psychological symptoms) that occurs during the luteal phase of the menstrual cycle. Dysmenorrhea is a sort of period pelvic pain, caused by blood flow decrease abruptly and ischemia due to frequent contraction of the uterus.

In clinical practice, gynecologists apply analgesic such as Non-steroidal Anti- inflammatory Drugs (NSAIDs), and oral contraceptive pills (OCT) or progestin as conventional therapy for premenstrual syndrome and dysmenorrhea. As NSAIDs may cause gastrointestinal discomfort, dyspepsia while hormone therapy leads to other concerns; some women now adopt acupuncture as an alternative therapy for its safety. However, many parameters affect the efficacy of acupuncture, such as the sorts of acupoints (of which meridians) or the numbers of acupoints; and proper evidence-based medicine on this issue is few.

Therefore, in this study, we aim to evaluate 1. The different impact of acupuncture and conventional therapy in premenstrual syndrome and dysmenorrhea women ; 2. Will the character (of which meridians) or numbers of acupoints be affecting factors of efficacy in treating premenstrual syndrome and dysmenorrhea? 3. Shall there be any relationship between the acupuncture and autonomic nerve activity adjustment in premenstrual syndrome and dysmenorrhea? 4. Shall there be any relationship between the acupuncture and TCM syndrome adjustment in premenstrual syndrome and dysmenorrhea?

DETAILED DESCRIPTION:
Subjects in this study included premenstrual syndrome and dysmenorrhea.

Premenstrual syndrome (PMS) is the sum of a group of symptoms (including physical and psychological symptoms) that occurs during the luteal phase of the menstrual cycle. Women who have such symptoms have been estimated as high as 75%; of which 3% to 8% are severe symptoms, called premenstrual dysphoric disorder (premenstrual dysphoric syndrome, PMDD). The two groups are very similar. Premenstrual syndrome is mostly for physical discomfort, while premenstrual dysphoric syndrome is for emotional problems, affecting women's sleep seriously.

Dysmenorrhea is a sort of period pelvic pain, caused by blood flow decrease abruptly and ischemia due to frequent contraction of the uterus. Many females afflicted with dysmenorrhea to different extents; some suffered from depression, reduced the quality of life; others even need to withdraw from work or school for incapable of daily activity. Thus, dysmenorrhea causes a lot of health burden and worth our attention. The prevalence of dysmenorrhea is up to 50 %. Generally speaking, primary dysmenorrhea is a menstrual pain in the absence of pelvic pathology while secondary dysmenorrhea is caused by organic dysfunction such as endometriosis, uterus malformation, cervix structure, pelvic inflammation, etc.

In clinical practice, gynecologists apply analgesic such as Non-steroidal Anti- inflammatory Drugs (NSAIDs), and oral contraceptive pills (OCT) or progestin as conventional therapy for premenstrual syndrome and dysmenorrhea. As NSAIDs may cause gastrointestinal discomfort, dyspepsia while hormone therapy leads to other concerns; some women now adopt acupuncture as an alternative therapy for its safety. However, many parameters affect the efficacy of acupuncture, such as the sorts of acupoints (of which meridians) or the numbers of acupoints; and proper evidence-based medicine on this issue is few. According to the theory of Traditional Chinese Medicine, acupuncture regulates meridians' energy and coordinates yin/yang while the western medicine reveals that the mechanism of pain-control of acupuncture is relevant to the theory of neurophysiology and some neuropeptide releasing, such as endorphin. Additionally, in our previous study, we noted that the theory of yin/yang (meridian) is compatible with autonomic nerve theory. Since many symptoms women with Premenstrual Syndrome and dysmenorrhea suffered, such as poor sleep, anxiety, convulsion of the uterine muscle, are related to autonomic nerve dysfunction, we are intrigued to know whether or not the effect of acupuncture relates to adjusting autonomic nerve system. Therefore, in this study, we aim to evaluate 1. The different impact of acupuncture and conventional therapy in premenstrual syndrome and dysmenorrhea women ; 2. Will the character (of which meridians) or numbers of acupoints be affecting factors of efficacy in treating premenstrual syndrome and dysmenorrhea? 3. Shall there be any relationship between the acupuncture and autonomic nerve activity adjustment in premenstrual syndrome and dysmenorrhea? 4. Shall there be any relationship between the acupuncture and TCM syndrome adjustment in premenstrual syndrome and dysmenorrhea? We expect through this multidisciplinary study; we can coordinate not only the different viewpoints of both Chinese and western medicine but also verify the compatibility of the theory of yin/yang and autonomic nerve (parasympathetic/sympathetic). We look forward the study can not only be a reference for further evidence-based research but also by reconciling different perspectives of Chinese and western medicine, we can, in turn, promote the cross-talk of Chinese and Western medicine in practical and academic aspects.

ELIGIBILITY:
Inclusion Criteria:

1. Women within reproductive age (15 to 49 years)
2. VAS≧4
3. Women with a history of regular menstrual cycles (28days±7 days)
4. Self-reported lower abdominal and pelvic, medial anterior thigh pain or low back pain associated with the onset of menses and lasting in 72 hours.

4.Symptoms: dysmenorrhagia, breast pain, dizziness, bloating, cramps, nausea, vomiting, diarrhea, headache, fatigue, etc.

Exclusion Criteria:

1. Women with irregular menstrual cycles
2. Women use of an intrauterine contraceptive device (IUCD/IUD)
3. Women with uncontrolled neurological diseases
4. Lactation, pregnant women, or those with plans to get pregnant in the coming half year

Ages: 19 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 105 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Wang Qi Chinese Medicine Questionnaire | We will evaluate separately at baseline and the end of cycle 4 (each cycle is 30 days). Change from Baseline TCM constitutions at 4 cycles (each cycle is 30 days). Time Frame: baseline and 4 cycles (each cycle is 30 days)
  This questionnaire is used to survey TCM constitutions. Evaluate body constitution of each individual by score(Balanced Constitution, Qi-deficient Constitution, Yang-deficient Constitution, Yin-deficient Constitution, Phlegm-dampness Constitution, Damp-heat Constitution, Stagnant Blood Constitution, Stagnant Qi Constitution, and Inherited Special Constitution).
Heart rate variation (HRV) test | We will evaluate separately at baseline and the end of cycle 4 (each cycle is 30 days). Change from Baseline HRV parameter at 4 cycles (each cycle is 30 days). Time Frame: baseline and 4 cycles (each cycle is 30 days)
  HRV test include time domain analysis and frequency domain analysis.Time domain analysis includes SDNN, R-MSSD and pNN50. Frequency domain analysis includes LF, HF, LF/HF and total power.

SECONDARY OUTCOMES:
Visual analogue scale(VAS) score | We will evaluate separately at baseline and the end of cycle 4 (each cycle is 30 days). Change from Baseline VAS score at 4 cycles (each cycle is 30 days). Time Frame: baseline and 4 cycles (each cycle is 30 days)
  VAS is used to assess the extent of menstrual pain.
Verbal multidimensional scoring system (VMSS) assessment | We will evaluate separately at baseline and the end of cycle 4 (each cycle is 30 days). Change from Baseline VMSS assessment at 4 cycles (each cycle is 30 days). Time Frame: baseline and 4 cycles (each cycle is 30 days)
  VMSS is used to assess the severity of dysmenorrhea. The VMSS assessment ranges from zero, one, two and three grade for evaluating the working ability, the systemic symptoms and whether analgesia is required or not.
  Grade 0 indicates that menstruation is not painful and daily activity is unaffected.
  Grade 1 indicates that menstruation is painful but seldom inhibits normal activity; analgesics are seldom required; mild pain.
  Grade 2 indicates that daily activity is affected; analgesics required and give sufficient relief so that absence from school is unusual; moderate pain.
  Grade 3 indicates that activity clearly inhibited; poor effect of analgesics; vegetative symptoms (headache, fatigue, vomiting, and diarrhea); severe pain.
SF-12 Health Survey | We will evaluate separately at baseline and the end of cycle 4 (each cycle is 30 days). Change from Baseline SF-12 Health Survey at 4 cycles (each cycle is 30 days). Time Frame: baseline and 4 cycles (each cycle is 30 days)
  SF-12 health survey is a questionnaire used to assess the quality of life of individuals. It contains a total of 12 questions and can be aggregated into physiological facets and psychological facets to assess the physiological and mental health status of the subjects.
Blood test | We will evaluate separately at baseline and the end of cycle 4 (each cycle is 30 days). Change from Baseline blood test at 4 cycles (each cycle is 30 days). Time Frame: baseline and 4 cycles (each cycle is 30 days)
  Contain:estrogen, progesterone and prostaglandin
Menstrual Distress Questionnaire(MDQ) | We will evaluate separately at baseline and the end of cycle 4 (each cycle is 30 days). Change from Baseline Menstrual Distress Questionnaire at 4 cycles (each cycle is 30 days). Time Frame: baseline and 4 cycles (each cycle is 30 days)
  Contain: Pain；Concentration；Behavioral Change；Autonomic Reactions；Water Retention；Negative Affect

CONTACTS AND LOCATIONS:
Overall Officials: Tsai-Ju Chien, PhD degree, Principal Investigator — Taipei City Hospital; Yi-Shuo Huang, B.S. degree, Study Director — Taipei City Hospital
Locations (1):
- Taipei City H, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
This study will have a continuous plan.